CLINICAL TRIAL: NCT02914093
Title: Feasibility of Inspiratory Muscle Training in Patients With Chronic Hypercapnia and Severe Chronic Obstructive Pulmonary Disease
Brief Title: IMT in Hypercapnic Patients With COPD
Acronym: THYPISK-f
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Linette Marie Kofod, Physiotherapist, Hvidovre University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-16022336
Record Dates: First submitted 2016-07-19; First posted 2016-09-26 (Estimated); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: COPD
Keywords: Hypercapnia; Physiotherapy; Inspiratory Muscle Training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypercapnia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IMT-feasibility (Experimental): Single arm intervention
  Interventions: Other: IMT

INTERVENTIONS:
Other: IMT — Inspiratory muscle training for 6 weeks 2x30 breaths daily as a home based program

SUMMARY:
The overall objective of the study is to investigate the feasibility of home based inspiratory muscle training (IMT) on chronic hypercapnia in patients with severe COPD, and to examine the relationship between inspiratory muscle strength and carbon dioxide level.

DETAILED DESCRIPTION:
The development of chronic hypercapnia in patients with COPD indicates an imbalance of increased ventilatory work caused by hyperinflation and airway resistance and a decreased inspiratory muscle reserve, probably caused by diaphragm- dysfunction. The inspiratory muscle strength can be trained by a devise, which provides a resistance to inspiration.

This study will be conducted as an a feasibility study and will examine whether inspiratory muscle training with a Power Breathe device (K3) is possible over a 6 week period in patients with COPD and chronic hypercapnia (pCO2 > 6 kilo pascal).

IMT will be considered as feasible if 80% of the planned training sessions have been completed, and if the maximum inspiratory strength improves by an average of 10% from MIP and if patients do not experience any discomfort or increased dyspnea during training.

The training of the respiratory strength is carried out daily with an electronic handheld device (Power Breathe K3) and will consist of 2x30 inspirations per day with the resistance adjusted individually and progressively with a pressure of 30 - 50% of maximal inspiratory pressure. Training will take place in the home.

ELIGIBILITY:
Inclusion Criteria:

* Have the diagnosis COPD with FEV1 / FVC <0.70 and FEV1 <50%
* Have elevated pCO2 in stable phase assessed by arterial blood gas with pCO2> 6 kPa
* Have given informed consent
* Can understand written and oral instructions

Exclusion Criteria:

* Patients are included in other projects with impact on the carbon dioxide level, e.g. home noninvasive ventilation treatment
* Patients using variable oxygenation rate that may affect the carbon dioxide level.
* Unstable patients and at high risk of exacerbation during the investigation period
* Hospitalized patient with COPD exacerbation during the intervention period
* Patients with an expected need for change of COPD medication or oxygen supply equipment in the study period.

The participation in the study will be postponed if the patient is in a rehabilitation program

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-09; Primary Completion 2018-05 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Completed training sessions | 6 weeks
  Feasibility - if 80% of the planned training sessions have been completed
Changes i Pimax | 6 weeks
  Feasibility - if the maximum inspiratory strength measured in cmH2O improves by an average of 10 %
Experienced discomfort | 6 weeks and during the training session
  Feasibility - if the patients do not experience any discomfort or increased dyspnea during and after training

SECONDARY OUTCOMES:
Changes in pCO2 | 6 weeks
  Arterial bloodgas analysis at day 1 and day 42 to measure pCO2 in kPa before and after the intervention
6 minutes walking test | 6 weeks
  6 MWT assess the distance walked over six minutes as a sub-maximal test of aerobic capacity/ endurance
CAT | 6 week
  CAT (COPD Assessment Test), symptom questionnaire, measured in points from 0- 40

CONTACTS AND LOCATIONS:
Overall Officials: Morten T Kristensen, PhD, Study Chair — Copenhagen University Hospital, Hvidovre; Ejvind F Hansen, MD, Study Chair — Pulmonary Sektion, Copenhagen University Hospital, Hvidovre
Locations (1):
- Copenhagen University Hospital, Hvidovre, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No